CLINICAL TRIAL: NCT01343446
Title: Sleep Impairment Can Influence The Coping Style Of Patients With Diabetes
Brief Title: Sleep Impairment and Coping Style in Diabetes
Acronym: Diabetesleep
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Istanbul University, Cerrahpasa School of Medicine
Other Study IDs: Cer-Met-A2
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Obesity; Sleep Disorders; Coping Skills
Keywords: Sleep impairment, Coping Style, Diabetes Mellitus
MeSH Terms: conditions — Obesity; Sleep Wake Disorders; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Diabetes: Patients with diabetes suffer from sleep impairment or not

SUMMARY:
To examine the effect of sleep impairment on coping style of patients with diabetes

DETAILED DESCRIPTION:
Abstract Objective: To examine the effect of sleep impairment on coping style of patients with diabetes Research Design and Methods: A total of 105 patients (40 male, 65 female) with diabetes mellitus were recruited from outpatient diabetic clinics in 2011 February. All patients were asked to fill the sociodemographic inquiry, Epworth Sleepiness Scale and Coping Style Inventory.

ELIGIBILITY:
Inclusion Criteria:

- Patients with diabetes longer than 6 months

Exclusion Criteria:

- Complications as a congestive heart failure, chronic renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Followed-up in Cerrahpasa Clinics of Diabetes Patients with diabetes Patients with/without diabetic complication Patients suffer from sleep impairment
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Coping style of Patients with Diabetes suffer from Sleep Disorder | Up to 1 week (Patients at follow-up)
  Patients with diabetes had filled the Epworth Sleepiness Scale and Coping styles ınventory

CONTACTS AND LOCATIONS:
Overall Officials: Murat Emül, Assoc.Prof., Study Director — Department of Psychiatry, Cerrahpasa School of Medicine
Locations (1):
- Diabetes and Metabolism Outpatients Clinic of Cerrahpasa School of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Luyckx K, Seiffge-Krenke I, Hampson SE. Glycemic control, coping, and internalizing and externalizing symptoms in adolescents with type 1 diabetes: a cross-lagged longitudinal approach. Diabetes Care. 2010 Jul;33(7):1424-9. doi: 10.2337/dc09-2017. Epub 2010 Mar 31. PMID 20357383